CLINICAL TRIAL: NCT00196014
Title: Evaluation of a Tool to Measure a Nurse's Individual Perception of Workload
Brief Title: Individual Workload Perception Scale - Revised (IWPS-R)
Acronym: IWPS-R
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Susan Teasley, Manager Patient Care Services, Children's Mercy Hospital Kansas City
Other Study IDs: 1989
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: Registered Nurses; Workload; Clinical staff nurses that are currently working

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to validate the psychometrics of the Individual Workload Perception Scale (IWPS).

DETAILED DESCRIPTION:
The purpose of this study is to validate the psychometrics of the Individual Workload Perception Scale (IWPS) designed to measure the perception of individual workloads of inpatient registered nurses.

ELIGIBILITY:
Inclusion Criteria:

* Nurses

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: LPNS and Registered Nurses
Sampling Method: Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2001-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen S Cox, RN, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States

REFERENCES:
- [Background] Cox KS, Anderson SC, Teasley SL, Sexton KA, Carroll CA. Nurses' work environment perceptions when employed in states with and without mandatory staffing ratios and/or mandatory staffing plans. Policy Polit Nurs Pract. 2005 Aug;6(3):191-7. doi: 10.1177/1527154405279091. PMID 16443974
- [Background] Lacey SR, Teasley SL, Henion JS, Cox KS, Bonura A, Brown J. Enhancing the work environment of staff nurses using targeted interventions of support. J Nurs Adm. 2008 Jul-Aug;38(7-8):336-40. doi: 10.1097/01.NNA.0000323942.04888.36. PMID 18690124
- [Background] Lacey SR, Teasley SL, Cox KS. Differences between pediatric registered nurses' perception of organizational support, intent to stay, workload, and overall satisfaction, and years employed as a nurse in magnet and non-magnet pediatric hospitals: implications for administrators. Nurs Adm Q. 2009 Jan-Mar;33(1):6-13. doi: 10.1097/01.NAQ.0000343342.24925.0c. PMID 19092517
- [Result] Cox KS, Teasley SL, Zeller RA, Lacey SR, Parsons L, Carroll CA, Ward-Smith P. Know staff's "intent to stay". Nurs Manage. 2006 Jan;37(1):13-5. doi: 10.1097/00006247-200601000-00004. No abstract available. PMID 16395045
- [Result] Cox KS, Teasley SL, Lacey SR, Carroll CA, Sexton KA. Work environment perceptions of pediatric nurses. J Pediatr Nurs. 2007 Feb;22(1):9-14. doi: 10.1016/j.pedn.2006.05.005. PMID 17234494
- [Result] Teasley SL, Sexton KA, Carroll CA, Cox KS, Riley M, Ferriell K. Improving work environment perceptions for nurses employed in a rural setting. J Rural Health. 2007 Spring;23(2):179-82. doi: 10.1111/j.1748-0361.2007.00087.x. PMID 17397376
- [Result] Lacey SR, Cox KS, Lorfing KC, Teasley SL, Carroll CA, Sexton K. Nursing support, workload, and intent to stay in Magnet, Magnet-aspiring, and non-Magnet hospitals. J Nurs Adm. 2007 Apr;37(4):199-205. doi: 10.1097/01.NNA.0000266839.61931.b6. PMID 17415107
- [Result] Sexton KA, Hunt CE, Cox KS, Teasley SL, Carroll CA. Differentiating the workplace needs of nurses by academic preparation and years in nursing. J Prof Nurs. 2008 Mar-Apr;24(2):105-8. doi: 10.1016/j.profnurs.2007.06.021. PMID 18358445